CLINICAL TRIAL: NCT02280174
Title: Effect of Linagliptin on Intestinal Triglyceride-rich-lipoprotein Metabolism in Type 2 Diabetic Patients
Brief Title: Effect of Linagliptin on TRL Metabolism
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Public Health, Argentina (Other Government)
Collaborators: Aix Marseille Université (Other); Instituto de Biología y Medicina Experimental, IBYME, Buenos Aires, Argentina (Unknown)
Responsible Party: Principal Investigator, MD/PhD Nogueira, Juan Patricio, MD/PhD, Ministry of Public Health, Argentina
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: IS000586
Record Dates: First submitted 2014-10-28; First posted 2014-10-31 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Type 2 Diabetes
Keywords: Apo B-48; TRL; Linagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug: linagliptin (Experimental): linagliptin 5 mg/d for 12 weeks
  Interventions: Drug: linagliptin
- Drug: standard treatment (No Intervention): sulfonylurea treatment for 12 weeks

INTERVENTIONS:
Drug: linagliptin — linagliptin 5 mg/d for12 weeks
  Other Names: Trajenta®
  Arms: Drug: linagliptin

SUMMARY:
Overproduction of intestinally derived triglyceride-rich lipoproteins (TRLs) (chylomicrons) has recently been described in type 2 diabetes (T2DM), as is known for hepaticTRL (very-low-density lipoprotein) production.

There is an interest in identifying therapies that would favourably influence postprandial concentrations of lipids in T2DM.

linagliptin is a potent and selective inhibitor of dipeptidyl peptidase IV (DPP-IV), and has been shown to reduce fasting and postprandial glucose levels in patients with type 2 diabetes mainly through incretin hormone-mediated improvements in islet function.

Although clinical studies to date indicate that fasting lipid levels are minimally affected by DPP-IV inhibitor treatment, animal studies suggested that DPP-IV inhibition reduce intestinal triglycerides (TG) absorption and apolipoprotein (apo) production and increased chylomicron catabolism. Interestingly, a recent study supporting this hypothesis showed that vildagliptin therapy was able to reduce postprandial intestinal TRL particles in patients with type 2 diabetes. Recently, it had reported that sitagliptin treatment significantly reduced plasma apoB-48 and TG concentrations in the postprandial state.

The action of DPP-IV inhibitors may be explained by insulin secretion or action of glucagon-like peptide (GLP-1) on metabolism of TRL.

Therefore, the present study was designed to examine the effects of linagliptin treatment (LT) vs standard treatment (ST) on the metabolism of TRL apoB-48 in patients with type 2 diabetes over a 12 weeks-period.

The investigators will study the patients in three different moments defined as: Time 0 (2 weeks before LT or ST, Time 1 (4 weeks after LT or ST), Time 2 (12 weeks after LT or ST). With areas under the curve (AUCs) of apoB48 in postprandial conditions.

DETAILED DESCRIPTION:
Uncontrolled type 2 Diabetes patients with HbA1c between 7 and 10% Patients must have received the maximum tolerated dose of metformin for at least 3 months before randomization. Patients will be randomised to receive linagliptin or standard therapy.

A total of seven study visits will be scheduled: at screening, at weeks -4, -2, 0, 4, 6, 12 and 24 week follow-up. During each visit, an endocrinologist will make the physical and metabolic assessment. Safety and tolerability data will be collected at screening and throughout the study, and includes incidence of serious and non serious adverse events (AEs) in linagliptin arms and standard arms. Clinical laboratory data, vital signs, and 12-lead electrocardiogram parameters at each visit, will be collected. The causal relationships between study drugs and AEs will be evaluated by the investigators at site. All drug-related AEs occurring during the study will be followed up until relieved or judged to be no longer clinically significant. Changes in body weight from baseline until week 12 will also be assessed. Hypoglycaemic event intensity will be defined as symptoms of hypoglycemia accompanied by a fingerstick glucose value of ≤ 50 mg/dl.

The investigators will study the patients in three different moments defined as: Time 0 (2 weeks before LT or ST), Time 1 (4 weeks after LT or ST), Time 2 (12 weeks after LT or ST). T1 show the direct effect (independent of metabolic changes) and T2 show indirect effect (depend of metabolic changes).

In each phase, following an overnight fast, an intravenous catheter will be inserted into a superficial vein in each forearm for blood sampling. After an overnight fast, subjects were admitted in the research unit for a 24-h period and received un isocaloric (900 kcal), mixed meals (75 g carbohydrates, 50 g fat (60% saturated), 35 g protein), at time points 7.00 a.m. (breakfast). Blood samples will drawn before and 2, 4, 6, 8, after the meal. The area under curve (AUC) and incremental AUC (IAUC) for postprandial variables will calculate in each phase.

In the morning after each phase study: basal (T0) and incretin conditions (T1 and T2), subjects will undergo hyperglycaemic clamp and hyperinsulinaemic clamp, successively. The insulin secretion rate and insulin sensitivity index will be measured during the last 30 minutes of the clamp, respectively in two arms of the study.

ELIGIBILITY:
Inclusion Criteria:

* Men from 40 to 65 years old. (excluding women because of hormonal changes in post menopause period could be influenced lipid parameters)
* Type 2 diabetes as defined by the American Diabetes Association.
* Body mass index between 25 and 40.0 kg/m².
* Baseline glycated hemoglobin A1c (HbA1c) between 7 and 10 %.
* Patients having received stable doses of metformin for at least 3 months before randomization.
* Non-smoker.
* Subject without cardiovascular events 6 months ago. (the treatment with lipid lowering agents and beta blockers in this condition could be perturbed the lipids parameters)
* Subject is informed and is consented.
* Plasma without severe dyslipidaemia: plasma triglyceride levels <4.51mmol/L (<400 mg/dl), plasma HDL levels >1.0 mmol/L (>40 mg/dl), LDL-cholesterol <5.10 mmol/L (<200 mg/dl).

Exclusion Criteria:

* Patients having received or being treated with pioglitazone, GLP-1 analogues, insulin or anti-obesity drugs (orlistat) within the past 3 months will be excluded
* Patients taking any other hypoglycemic agent, other than metformin.
* Patients with type 1 diabetes, secondary diabetes or acute metabolic diabetic complications will be excluded.
* Subjects will be excluded if they have cardiovascular disease (coronary heart disease, cerebrovascular disease or peripheral arterial disease) or if they are taking other medications known to affect lipoprotein metabolism (e.g. steroids, beta blockers, thiazide diuretics, lipid lowering agents: (statins, fibrates, ezetimibe, niacin), significant alcohol intake etc.).
* Subjects who are in a situation or have any condition that, in the opinion of the investigator, may interfere with optimal participation in the study.
* Individuals with a history of mental instability, individuals who have been treated or are being treated for severe psychiatric illness that, in the opinion of the investigator, may interfere with optimal participation in the study.
* History of alcohol or drug abuse within the past 2 years. Patients must not take alcohol during the study.
* Disorders of the hematologic, digestive, or central nervous systems, including cerebrovascular disease and degenerative disease, that would limit study evaluation or participation.
* Known impairment of renal function (serum creatinine levels > 1.7 mg/dL for men), dysproteinemia, nephrotic syndrome, or other renal disease (24-hour urinary protein ≥3 ± 1 g).
* Active or chronic hepatobiliary or hepatic disease. In addition, patients with aspartate aminotransferase or alanine aminotransferase >2 x upper limit of the laboratory reference range will be excluded.
* Subjects with coagulopathy, prothrombin time (PT) or partial thromboplastin time (PTT) at Visit 1 >1.5 times control.
* Subjects with hemoglobin >2 x the lower limit of the laboratory reference range will be excluded.
* Patients who are known to have tested positive for human immunodeficiency virus (HIV).
* Patients who are currently enrolled in another clinical study.
* Patients who have used any investigational drug within 30 days of the first clinic visit.
* Congestive heart failure New York Heart Association (NYHA) Class III or IV. Uncontrolled cardiac arrhythmias within 3 months of study entry.
* Other endocrine or metabolic disease known to influence serum lipids or lipoproteins.
* known hypersensitivity or allergy to linagliptin or its excipients, metformin
* Unwillingness or language barrier precluding adequate understanding or cooperation.

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Measurement of the Area Under the Curve of Plasma apoB-48 Levels During Postprandial Period (Time 0,2,4,6,8 Hours) | At the end of the 12-week interventions

CONTACTS AND LOCATIONS:
Overall Officials: Juan Nogueira, MD/PhD, Principal Investigator — Medico Moving Center Institute, Formosa, Argentina
Locations (1):
- National University of Formosa, Formosa, Formosa Province, Argentina